CLINICAL TRIAL: NCT01346696
Title: An Open, Prospective, Multi-center Study Assessing the OsseoSpeed™ TX Length 6 mm in in the Posterior Maxilla and Mandible. A 3-years Follow-up Study.
Brief Title: Study on OsseoSpeed™ TX Short Implants in a Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-0005
Record Dates: First submitted 2011-05-02; First posted 2011-05-03 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Partially Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous, Partially

ARMS (1):
- OsseoSpeed™ TX implants (Experimental): OsseoSpeed TX implants; Ø 4.0 mm, length 6 mm.
  Interventions: Device: OsseoSpeed™ TX implant (Ø 4.0 mm, length 6 mm)

INTERVENTIONS:
Device: OsseoSpeed™ TX implant (Ø 4.0 mm, length 6 mm)

SUMMARY:
The purpose of this study is to investigate the clinical efficacy of OsseoSpeed™ TX 6 mm implants in a Chinese population by evaluation of marginal bone level alteration, implant stability and implant survival in the posterior mandible and maxilla up to 3 years after loading. The hypothesis is that one stage surgery using 6 mm OsseoSpeed™ TX implant in the posterior region is safe and predictable.

ELIGIBILITY:
Inclusion criteria:

1. Provision of informed consent
2. Female and male aged 20-75 years at enrolment
3. In need for 2-3 implants in either side of the posterior mandible or maxilla (premolar and molar region)
4. History of edentulism in the study area of at least four months
5. Neighboring tooth/teeth to the planned bridge/crowns must have natural root(s)
6. Presence of natural teeth, partial prosthesis and/or implants in the opposite jaw in contact with the planned bridge/crowns
7. Deemed by the investigator to be suitable for implants of 6 mm length and to have a bone height of at least 6 mm and a bone width of minimum 6 mm
8. Deemed by the investigator as likely to present an initially stable implant situation

Exclusion criteria:

1. Unlikely to be able to comply with study procedures, as judged by the investigator
2. Earlier graft procedures in the study area
3. Uncontrolled pathologic processes in the oral cavity
4. Known or suspected current malignancy
5. History of radiation therapy in the head and neck region
6. History of chemotherapy within 5 years prior to surgery
7. Systemic or local disease or condition that could compromise post-operative healing and/or osseointegration
8. Uncontrolled diabetes mellitus
9. Corticosteroids or any other medication that could influence post-operative healing and/or osseointegration
10. Smoking more than 10 cigarettes/day
11. Present alcohol and/or drug abuse
12. Involvement in the planning and conduct of the study (applies to both Astra Tech staff and staff at the study site)
13. Previous enrolment in the present study
14. Simultaneous participation in another clinical study, or participation in a clinical study during the last 6 months
15. Subjects that are unable to give informed consent

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huan Xin Meng, Prof, Principal Investigator — Department of Periodontology, School of Stomatology, Beijing University
Locations (3):
- China (3):
  - Department of Periodontology, School of Stomatology, Peking University, Beijing
  - Department of Implantology, School of Stomatology, Peking University, Beijing
  - Second Dental and Periodontal Center, School of Stomatology, Peking University, Beijing

REFERENCES:
- [Result] Han J, Zhang X, Tang Z, Zhang L, Shi D, Meng H. A prospective, multicenter study assessing the DENTSPLY Implants, OsseoSpeed() TX, length 6 mm in the posterior maxilla and mandible: a 1-year follow-up study. Clin Oral Implants Res. 2016 Apr;27(4):452-7. doi: 10.1111/clr.12587. Epub 2015 Apr 9. PMID 25855871
- [Result] Han J, Tang Z, Zhang X, Meng H. A prospective, multi-center study assessing early loading with short implants in posterior regions. A 3-year post-loading follow-up study. Clin Implant Dent Relat Res. 2018 Feb;20(1):34-42. doi: 10.1111/cid.12568. Epub 2017 Dec 8. PMID 29218810

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implants
Period: Overall Study
Arm/Group | OsseoSpeed™ TX Implants
Started | 45; 94 Implants
Completed | 44; 90 Implants
Not Completed | 1; 4 Implants
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX Implants
Number analyzed (Participants) | 45
Number analyzed (Implants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 17
Region of Enrollment [Number; unit: participants]
  China | 45

OUTCOME MEASURES:

1. Primary Outcome: Marginal Bone Level Alteration
Description: Marginal Bone Level determined from radiographs and expressed as the difference from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant, and expressed in millimeters. Marginal Bone Level change calculated from values obtained at delivery of permanent restoration i.e. loading of implants (baseline) compared to the values obtained at the follow-up visit 12 months after loading.
  Positive value = bone gain, Negative values = bone loss.
Time Frame: Evaluated from implant installation to 12 months after implant loading
Population: 45 subjects (90 implants) completed the 12-month follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 36 subjects (75 implants).
  Six of the collected radiographs were not possible to evaluate, giving an overall number of 35 subjects (69 implants) as basis for the 12 months analysis of MBL change.
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX Implants
Number analyzed (Participants) | 34
Number analyzed (Implants) | 69
millimeter | -0.06 (0.55)

2. Secondary Outcome: Marginal Bone Level Alteration After 36 Months
Description: Marginal Bone Level determined from radiographs and expressed as the difference from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant, and expressed in millimeters. Marginal Bone Level change calculated from values obtained at delivery of permanent restoration i.e. loading of implants (baseline) compared to the values obtained at the follow-up visit 36 months after loading.
  Positive value = bone gain, Negative values = bone loss.
Time Frame: Evaluated from implant loading to 36 months after implant loading.
Population: 44 subjects (90 implants) completed the 36-month follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 36 subjects (75 implants).
  Four of the collected radiographs were not possible to evaluate, giving an overall number of 35 subjects (71 implants) as basis for the 36 months analysis.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | OsseoSpeed™ TX Implants
Number analyzed (Participants) | 35
millimeter | 0.07 (0.49)

3. Secondary Outcome: Implant Survival
Description: Implant survival rate evaluated clinically and radiographically.
Time Frame: Evaluated from implant installation to 36 months after implant loading.
Population: 44 subjects (90 implants) completed the 36-month follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 36 subjects (75 implants).
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX Implants
Number analyzed (Participants) | 36
Number analyzed (Implants) | 75
Implants | 75

4. Secondary Outcome: Implant Stability
Description: Implant stability evaluated clinically/manually (recorded as stable yes/no).
Time Frame: Evaluated 36 months after implant loading.
Population: as for outcome 3
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX Implants
Number analyzed (Participants) | 36
Number analyzed (Implants) | 75
Implants | 75

5. Secondary Outcome: Condition of the Periimplant Mucosa (PPD).
Description: Condition of the periimplant mucosa measured by assessment of probing pocket depth (PPD).
  Change in pocket depth expressed in millimeters at the 36 month follow-up visit compared to values obtained at delivery of permanent restoration i.e. loading (baseline).
  Negative value = increased pocket depth
Time Frame: Evaluated from implant loading to 36 months after implant loading.
Population: 44 subjects (90 implants) completed the 36-month follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 36 subjects (75 implants).
  Baseline and/or follow-up measurements not available for 3 implants, giving an overall number of 36 subjects (72 implants) as basis for the 36 months analysis of PPD change.
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX Implants
Number analyzed (Participants) | 36
Number analyzed (Implants) | 72
millimeter | -0.63 (0.83)

6. Secondary Outcome: Condition of the Periimplant Mucosa (BoP).
Description: Condition of the periimplant mucosa will be measured by assessment of bleeding on probing (BoP).
  Presented as % of the implants that show presence of bleeding at time of the 36 months follow-up.
Time Frame: Evaluated from implant loading to 36 months after implant loading.
Population: 44 subjects (90 implants) completed the 36-month follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 36 subjects (75 implants).
  The BoP measurement was not completed for one implant, giving an overall number of 36 subjects (74 implants) as basis for the 36 months analysis of BoP.
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX Implants
Number analyzed (Participants) | 36
Number analyzed (Implants) | 74
Implants | 43

7. Secondary Outcome: Plaque
Description: Occurence of plaque around the study implant. Presented as proportion of implants that showed presence of plaque at the 36 months follow-up visit.
Time Frame: Evaluated 36 months after implant loading.
Population: 44 subjects (90 implants) completed the 36-month follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 36 subjects (75 implants).
  Plaque measurement was not completed for one implant, giving an overall number of 36 subjects (74 implants) as basis for the 36 months analysis of Plaque.
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX Implants
Number analyzed (Participants) | 36
Number analyzed (Implants) | 74
Implants | 29

8. Secondary Outcome: Crown-to-implant Ratio
Description: Crown height measured radiographically from the implant-abutment interface to the most coronal point on the prosthesis. The crown-to-implant ratio calculated from radiographs
Time Frame: 12 months after implant loading
Population: 45 subjects (90 implants) completed the 12-month follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 36 subjects (75 implants).
  6 of the collected radiographs were not possible to evaluate, giving an overall number of 35 subjects (68 implants) as basis for 12 months analysis of Crown-to-implant ratio.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX Implants
Number analyzed (Participants) | 35
Number analyzed (Implants) | 68
Ratio | 1.70 (0.32)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | OsseoSpeed™ TX Implants
Serious Adverse Events (participants affected / at risk) | 3/45
Other Adverse Events (participants affected / at risk) | 6/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsseoSpeed™ TX Implants (N=45)
Right femoral neck fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Hepatic hilum cholangiocarcinoma (Hepatobiliary disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsseoSpeed™ TX Implants (N=45)
Study implant not stable - implant lost (Investigations) | 4 (4) — 4 subjects lost one of their implants due to insufficient osseointegration. Those were all lost during the healing phase, before loading of the implant.
Study implant not stable - extended healing time (Investigations) | 3 (3) — 3 subjects had implants that required extended healing time in order to achieve stability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less